CLINICAL TRIAL: NCT02860364
Title: A Randomized Controlled Trial of Mild vs. Moderate Hypothermia on Patient Outcomes in Aortic Hemiarch Surgery With Anterograde Cerebral Perfusion
Brief Title: Comparing Hypothermic Temperatures During Hemiarch Surgery
Acronym: TITAN:COMMENCE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20160408
Record Dates: First submitted 2016-08-04; First posted 2016-08-09 (Estimated); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Thoracic Aortic Disease
MeSH Terms: interventions — Circulatory Arrest, Deep Hypothermia Induced

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mild Hypothermic Circulatory Arrest (Experimental): During aortic hemiarch surgery, mild hypothermia (32°C) will be used during circulatory arrest.
  Interventions: Procedure: Hypothermic circulatory arrest
- Moderate Hypothermic Circulatory Arrest (Active Comparator): During aortic hemiarch surgery, moderate hypothermia (26°C) will be used during circulatory arrest.
  Interventions: Procedure: Hypothermic circulatory arrest

INTERVENTIONS:
Procedure: Hypothermic circulatory arrest — During cardiac surgery requiring circulatory arrest, the patient's body temperature is lowered significantly to reduce the cellular metabolic rate and reduce ischemic injury.

SUMMARY:
Hypothermic circulatory arrest is an important surgical technique, allowing complex aortic surgeries to be performed safely. Hypothermic circulatory arrest provides protection to cerebral and visceral organs, but may result in longer cardiopulmonary bypass times during surgery, increased risks of bleeding, inflammation, and neuronal injury. To manage these consequences, a trend towards warmer core body temperatures during circulatory arrest has emerged. This trial will randomize patients to either mild (32°C) or moderate (26°C) hypothermia during aortic hemiarch surgery to determine if mild hypothermia reduces the length of cardiopulmonary bypass time and other key measures of morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Elective aortic hemiarch surgery
* Planned unilateral selective anterograde cardioplegia
* Anticipated lower body arrest time of < 20 minutes
* Able to provide written informed consent

Exclusion Criteria:

* Surgery for acute aortic dissection or emergent operations
* Total arch replacement
* Inability to perform unilateral selective anterograde cerebral perfusion (uSACP)
* Patients with known/documented coagulopathy
* Patients with cold agglutinin disease or those that test positive on routine preop screening
* Pre-existing severe neurological impairment or inability to accurately assess neurocognitive function as determined by the operating surgeon
* Severe carotid disease, defined as: any patient with previously documented carotid stenosis of > 70% (via Doppler ultrasound (US), magnetic resonance angiography (MRA), or computer tomography angiography (CTA)) without neurological deficits; or carotid stenosis > 50% with neurological deficits; or previous carotid endarterectomy or stenting
* Patients in renal failure or currently being treated with renal replacement therapy (RRT) or estimated glomerular filtration rate (eGFR) < 30 ml/min/1.73m2
* Use of an investigational drug or device at time of enrollment
* Participation in another clinical trial which interferes with performance of the study procedures or assessment of the outcomes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Estimated)
Dates: Start 2018-02-20 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Composite endpoint of neurologic and acute kidney injury | Up to 90 days after surgery.
  The primary objective of this study is to determine whether mild hypothermia (32°C) during aortic hemiarch surgery using unilateral selective anterograde cerebral perfusion (uSACP), is superior to moderate hypothermia (26°C) in reducing the composite endpoint of neurologic and acute kidney injury.

SECONDARY OUTCOMES:
Rates of Neurologic Injury | Up to 90 days after surgery.
  Comparison of mild (32°C) vs moderate (26°C) hypothermia in aortic hemiarch surgery with respect to incidence of neurologic injury, including transient ischemic attack (TIA) and permanent neurological dysfunction (PND) or stroke.
Incidence of Silent Strokes | Up to 90 days after surgery.
  Comparison of mild (32°C) vs moderate (26°C) hypothermia in aortic hemiarch surgery with respect to the incidence of silent strokes, defined as infarctions identified during magnetic resonance imaging (MRI) in patients without neurologic symptoms.
Incidence of Acute Kidney Injury (AKI) | Up to 90 days after surgery.
  Comparison of mild (32°C) vs moderate (26°C) hypothermia in aortic hemiarch surgery with respect to the incidence of acute kidney injury (AKI), defined as Stage 1 or greater using the KDIGO criteria. Using the KDIGO criteria, Stage 1 AKI is defined as an increase in serum creatinine of 1.5-1.9x the baseline or an increase >= 27umol/L with urine output <0.5mL/kg/hour for 6-12 hours.
Incidence of Delirium | Up to 90 days after surgery.
  Comparison of mild (32°C) vs moderate (26°C) hypothermia in aortic hemiarch surgery with respect to the incidence of delirium, using the Confusion Assessment Method (CAM). The Confusion Assessment Method defines delirium as the presence of acute changes in mental status with fluctuating course, plus inattention and the presence of either disorganized thinking OR altered level of consciousness.
Death | Up to 90 days after surgery.
  Comparison of mild (32°C) vs moderate (26°C) hypothermia in aortic hemiarch surgery with respect to the incidence of death
Evaluate differences in the duration of cardiopulmonary bypass used in patients who receive mild or moderate hypothermic circulatory arrest during aortic hemiarch surgery | During the index procedure
  Comparison of mild (32°C) vs moderate (26°C) hypothermia in aortic hemiarch surgery with respect to the length of time that the patient remains on cardiopulmonary bypass.
Rates of Mediastinal re-exploration for bleeding | Up to 90 days after surgery.
  Comparison of mild (32°C) vs moderate (26°C) hypothermia in aortic hemiarch surgery with respect to the rates of mediastinal re-exploration (re-operation) for bleeding.
Incidence and quantity of perioperative blood transfusions | Up to 90 days after surgery.
  Comparison of mild (32°C) vs moderate (26°C) hypothermia in aortic hemiarch surgery with respect to the number and quantity of perioperative blood transfusions
Incidence of prolonged Mechanical Ventilation | Up to 90 days after surgery.
  Comparison of mild (32°C) vs moderate (26°C) hypothermia in aortic hemiarch surgery with respect to the duration of mechanical ventilation. Mechanical ventilation will be defined as use of a mechanical ventilator ≥48 hours.
Perioperative Myocardial Infarction | Up to 48 hours after surgery.
  Comparison of mild (32°C) vs moderate (26°C) hypothermia in aortic hemiarch surgery with respect to the incidence of perioperative myocardial infarction. This will be clinically diagnosed using a combination of electrocardiographic (new Q wave on 12 lead ECG) and/or biochemical (TnI > 45 ng/L) markers.
Length of Stay | Up to 90 days after surgery.
  Comparison of mild (32°C) vs moderate (26°C) hypothermia in aortic hemiarch surgery with respect to the duration of a patient's stay in the intensive care unit and on the hospital ward.
Quality of life (SF-12) | Up to 90 days after surgery.
  Comparison of mild (32°C) vs moderate (26°C) hypothermia in aortic hemiarch surgery with respect to the patient's quality of life measured using the Short Form (SF) 12 questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Munir Boodhwani, MD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (12):
- United States (3):
  - Massachusetts General, Boston, Massachusetts
  - The Valley Hospital, Ridgewood, New Jersey
  - Ohio State University Medical Center, Columbus, Ohio
- Canada (9):
  - Kelowna General Hospital, Kelowna, British Columbia
  - Fraser Health Authority, Surrey, British Columbia
  - University of British Columbia, Vancouver, British Columbia
  - Dalhousie university, Halifax, Nova Scotia
  - London Health Sciences Centre, London, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - University Health Network, Toronto, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - Institut universitaire de cardiologie et de pneumologie de Québec, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made available to other researchers.

REFERENCES:
- [Derived] Jabagi H, Wells G, Boodhwani M. COMMENCE trial (Comparing hypOtherMic teMperaturEs duriNg hemiarCh surgEry): a randomized controlled trial of mild vs moderate hypothermia on patient outcomes in aortic hemiarch surgery with anterograde cerebral perfusion. Trials. 2019 Dec 9;20(1):691. doi: 10.1186/s13063-019-3713-9. PMID 31815641